CLINICAL TRIAL: NCT01126177
Title: A Randomised, Double-blind, Placebo-controlled Phase II Study, Comparing the Efficacy and Safety of Inhaled SNG001 to Placebo Administered to Asthmatic Subjects After the Onset of a Respiratory Viral Infection for the Prevention or Attenuation of Asthma Symptoms Caused by Respiratory Viruses
Brief Title: Comparing Efficacy and Safety of Inhaled SNG001 to Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synairgen Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG005
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo once daily for 14 days
  Interventions: Drug: Placebo
- SNG001 (Experimental)
  Interventions: Drug: Interferon beta 1a

INTERVENTIONS:
Drug: Interferon beta 1a — SNG001, IFN-β1a solution for inhalation
  Arms: SNG001
Drug: Placebo — Placebo (excipients of the SNG001 solution only)
  Arms: Placebo

SUMMARY:
When people with asthma get respiratory virus such as a cold or flu it often increases asthma symptoms. The investigators will test the study medication to find out if it can prevent the virus spreading from the nose to the lungs.

SNG001 contains Interferon-beta that occurs naturally in the body. In this study, SNG001 will be given by a nebuliser.

DETAILED DESCRIPTION:
The study will consist of a Pre-Treatment Phase into which subjects potentially eligible for the Treatment Phase will be recruited. Subjects will remain in the Pre-Treatment Phase until they experience respiratory virus symptoms at which time they will be further screened for eligibility for entry into the Treatment Phase. If eligible, subjects will be randomised 1:1 to receive SNG001 or placebo once daily for 14 days. Doses will be delivered by a CE marked breath actuated nebuliser (I-neb Philips Respironics). Subjects will be assessed for changes in changes in respiratory virus symptoms and asthma symptoms at home using a text message system, and via telephone questionnaire. Lung function will be measured both at home by the subjects (PEFR only) and in the clinic. Efficacy and safety will be monitored until at least 30 days post treatment.

ELIGIBILITY:
1. Male or female aged 18 to 65 years of age at the time of screening.
2. Symptoms of asthma for at least 2 years pri or to the Screening Visit, confirmed by a medical history and:

   1. ≥12% and 200mL bronchodilator reversibility at screening or documented in the past, OR,
   2. evidence of bronchial hyper-responsiveness at screening or documented in the past, OR,
   3. a documented hospital admission (including an Accident and Emergency admission) for asthma since the age of 18, OR.
   4. documented evidence that they have attended their GP surgery, out-of-hours clinic (or alternative health care provider) for worsening of asthma symptoms, since the age of 18
3. Must answer "Yes" to the question "Does a cold make your asthma worse?"
4. To have had at least one asthma exacerbation suspected to have been caused by a respiratory virus in the last 24 months which required the use of oral steroids and/or additional treatment with antibiotics on one or more occasion.
5. Must be taking regular inhaled corticosteroids.
6. Pre-bronchodilator FEV1 ≥ 40 % predicted at screening.
7. Post-bronchodilator FEV1 ≥ 50 % predicted at screening.
8. Provide written informed consent.
9. Females of childbearing potential must be using a medically acceptable adequate form of birth control and agree to maintain this usage throughout the duration of and four weeks post the Treatment Phase of the study.
10. Motivation (in the Investigator"s opinion) to complete all study visits, the ability to communicate well with the Investigator and be capable of understanding the nature of the research and its treatment including its risks and benefits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
S-ACQ | Baseline - Day 8
  To evaluate the superiority of inhaled SNG001 compared to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of asthma symptoms caused by respiratory viruses in the modified intention to treat (mITT) population as measured by change from Baseline to Day 8 in the Shortened-Asthma Control Questionnaire (symptoms plus short-acting β2 agonist.
  - change from Baseline to Day 8 in the Shortened-Asthma Control Questionnaire

SECONDARY OUTCOMES:
Asthma Index | Day 1-14
  To evaluate the superiority of inhaled SNG001 compared to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of asthma symptoms caused by respiratory viruses in the mITT population as measured by peak score of the Asthma Index (Sorkness et al, 2008) in the 14 day period following first administration of study drug (measured from 24 hours post first dose to 24 hours post last dose taken).
S-ACQ | Baseline - Day 8
  To evaluate the superiority of inhaled SNG001 compared to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of asthma symptoms caused by respiratory viruses in the per protocol (PP) population as measured by change from Baseline to Day 8 in the Shortened-Asthma Control Questionnaire.
Asthma Index | 14 days
  To evaluate the superiority of inhaled SNG001 compared to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of asthma symptoms caused by respiratory viruses in the PP population as measured by peak score of the Asthma Index in the 14 day period following first administration of study drug (measured from 24 hours post first dose to 24 hours post last dose taken).
Sever Exacerbation | Day 1-14
  To evaluate the superiority of inhaled SNG001 compared to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of asthma symptoms caused by respiratory viruses as measured by the proportion of subjects experiencing a severe exacerbation (Appendix 2) in the mITT population during the 14 days following first administration of study drug.
Lung Function | Day 1-14
  To compare inhaled SNG001 to placebo administered to asthmatic subjects after the onset of a respiratory viral infection for the prevention or attenuation of decreases in lung function (AUC FEV1 and PEFR) caused by respiratory viruses in the mITT population during the 14 day dosing period.
Viral Load | Days 4 and 7
  To compare the effect of inhaled SNG001 to placebo when administered to asthmatic subjects on viral load on Days 4 and 7 in sputum.
Safety | Day 1-14
  To evaluate the safety of inhaled SNG001 when administered to asthmatic subjects.
Concomitant Medications | Day 1-28
  To compare the frequency of use of concomitant medications in relation to conditions of the respiratory tract during the study Treatment Phase in asthmatic subjects receiving inhaled SNG001 compared to placebo.
Pharmacokinetic | Day 1-14
  To gain information on the pharmacokinetic profile of inhaled SNG001 administered to asthmatic subjects during a respiratory virus infection.
Pharmacodynamic | Day 1-14
  To gain information on the pharmacodynamic profile of inhaled SNG001 administered to asthmatic subjects during a respiratory virus infection.

CONTACTS AND LOCATIONS:
Overall Officials: Ratko Djukanovic, MD, DM, FRCP, Principal Investigator — University of Southampton
Locations (1):
- Southampton University General Hospital, Southampton, Hampshire, United Kingdom

REFERENCES:
- [Derived] Djukanovic R, Harrison T, Johnston SL, Gabbay F, Wark P, Thomson NC, Niven R, Singh D, Reddel HK, Davies DE, Marsden R, Boxall C, Dudley S, Plagnol V, Holgate ST, Monk P; INTERCIA Study Group. The effect of inhaled IFN-beta on worsening of asthma symptoms caused by viral infections. A randomized trial. Am J Respir Crit Care Med. 2014 Jul 15;190(2):145-54. doi: 10.1164/rccm.201312-2235OC. PMID 24937476